CLINICAL TRIAL: NCT04235920
Title: Correlation of Alberta Stroke Program Early CT Score (ASPECTS) With Cognitive Impairment and Outcome of Acute Ischemic Stroke
Brief Title: Cognitive Impairment and Outcome of Acute Ischemic Stroke.
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University 12
Record Dates: First submitted 2020-01-17; First posted 2020-01-22 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Stroke; Cognitive Impairment; Outcome, Fatal
Keywords: Stroke; ASPEACTS, Modified Rankin Scale, National Institutes of Health Stroke Scale. Higher cortical functions, Biomarkers of cognitive impairment.
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Impaired Cognition: First group was cognitively impaired test with MoCA score of 25 or less.
  Interventions: Diagnostic Test: Montreal Cognitive Assessment (MoCA)
- Preserved cognition: The second group was cognitively preserved with MoCA score of higher than 25.
  Interventions: Diagnostic Test: Montreal Cognitive Assessment (MoCA)

INTERVENTIONS:
Diagnostic Test: Montreal Cognitive Assessment (MoCA) — This scale evaluates different domains of cognition like attention, orientation, memory, language, visuoconstructional capacities, and lastly, executive functions. MoCA is a thirty point test with a score of 25 or less considered as abnormal impaired cognition

SUMMARY:
The aim of this study is to assess the use of ASPECTS and stroke biomarkers to predict the outcome and cognitive impairment in acute ischemic stroke.

DETAILED DESCRIPTION:
150 patients (79 males, and 71 females with a mean age of 64.05±11.55 years) were included in this study presented by acute middle cerebral artery territory ischemic stroke. Vascular risk factors were determined from the history taking. Assessment of GCS and NIHSS at the initial presentation was done to assess the stroke severity. Cognitive functions were evaluated in all study participants by the Montreal Cognitive Assessment (MoCA) Arabic version. An initial and follow up non-contrast CT brain was done after 7 days which were assessed by ASPECTS. Functional outcomes in stroke cases were assessed after three months by Glasgow Coma Scale, National Institutes of Health Stroke Scale and modified Rankin Scale. Biomarkers of cognitive impairment like ESR, CRP, S100B, MMP9 and glutamate were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* First attack of acute MCA territory infarction within 2 days from the onset.

Exclusion Criteria:

* previous stroke,
* presence of anterior cerebral artery infarction,
* posterior cerebral artery infarction, and
* venous infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 79 males and 71 females with a mean age of 64.05 ±11.55 were included in this study and were admitted with the first attack of acute MCA territory infarction within 2 days from the onset and aged more than 18 years. Acute ischemic stroke (AIS) was defined as a rapidly developing neurological deficit with an obvious known onset, and an initial CT brain with no proof of ICH.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 3 month after discharge
  This scale evaluates different domains of cognition like attention, orientation, memory, language, visuoconstructional capacities, and lastly, executive functions. MoCA is a thirty point test with a score of 25 or less considered as abnormal impaired cognition
Assessment of CT brain was done by ASPECTS. | 7 days
  The ASPECTS scoring was calculated for all patients. CT brain images were assessed for proof of localized parenchymal hypo-attenuation, loss of differentiation between gray and white matter, and if there is effacement of sulci. ASPECTS gives reliable methods for evaluation of ischemic stroke by utilizing a ten-point score "M1, M2, M3, M4, M5, M6, I: insula, IC: internal capsule, L: lentiform, and C: caudate" everyone represents one point. A Score of 10 means a normal CT scan. One point is decreased for each affected area on the CT brain. So, a score of 0 indicates widespread ischemia affecting the MCA territory

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mokin M, Primiani CT, Siddiqui AH, Turk AS. ASPECTS (Alberta Stroke Program Early CT Score) Measurement Using Hounsfield Unit Values When Selecting Patients for Stroke Thrombectomy. Stroke. 2017 Jun;48(6):1574-1579. doi: 10.1161/STROKEAHA.117.016745. Epub 2017 May 9. PMID 28487329
- [Background] Taylor-Rowan M, Wilson A, Dawson J, Quinn TJ. Functional Assessment for Acute Stroke Trials: Properties, Analysis, and Application. Front Neurol. 2018 Mar 26;9:191. doi: 10.3389/fneur.2018.00191. eCollection 2018. PMID 29632511
- [Background] Schroder J, Cheng B, Ebinger M, Kohrmann M, Wu O, Kang DW, Liebeskind DS, Tourdias T, Singer OC, Christensen S, Campbell B, Luby M, Warach S, Fiehler J, Fiebach JB, Gerloff C, Thomalla G; STIR and VISTA Imaging Investigators. Validity of acute stroke lesion volume estimation by diffusion-weighted imaging-Alberta Stroke Program Early Computed Tomographic Score depends on lesion location in 496 patients with middle cerebral artery stroke. Stroke. 2014 Dec;45(12):3583-8. doi: 10.1161/STROKEAHA.114.006694. Epub 2014 Oct 14. PMID 25316278
- [Background] Tan JP, Li N, Gao J, Wang LN, Zhao YM, Yu BC, Du W, Zhang WJ, Cui LQ, Wang QS, Li JJ, Yang JS, Yu JM, Xia XN, Zhou PY. Optimal cutoff scores for dementia and mild cognitive impairment of the Montreal Cognitive Assessment among elderly and oldest-old Chinese population. J Alzheimers Dis. 2015;43(4):1403-12. doi: 10.3233/JAD-141278. PMID 25147113
- [Derived] Esmael A, Elsherief M, Eltoukhy K. Predictive Value of the Alberta Stroke Program Early CT Score (ASPECTS) in the Outcome of the Acute Ischemic Stroke and Its Correlation with Stroke Subtypes, NIHSS, and Cognitive Impairment. Stroke Res Treat. 2021 Jan 29;2021:5935170. doi: 10.1155/2021/5935170. eCollection 2021. PMID 33575025